CLINICAL TRIAL: NCT03681223
Title: A Prospective Randomized Trial Comparing Restorelle® Y Mesh vs. Vertessa® Lite Y Mesh for Laparoscopic and Robotic-assisted Laparoscopic Sacrocolpopexy
Brief Title: Restorelle® Y Mesh vs. Vertessa® Lite Y Mesh for Laparoscopic and Robotic-assisted Laparoscopic Sacrocolpopexy
Acronym: Lite-Y
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-907
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Vaginal Vault Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: All subjects will be predetermined by their surgeon to undergo either a laparoscopic or robotic assisted laparoscopic sacrocolpopexy depending upon their clinical evaluation. The participants will then be randomized to either Restorelle® or Vertessa® Y sacrocolpopexy according to a computer-generated randomization.
Who Masked: Participant
Masking Description: All patients will be blinded to their assignment, investigators will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Restorelle® Y mesh (Active Comparator): All subjects will be predetermined by their surgeon to undergo either a laparoscopic or robotic assisted laparoscopic sacrocolpopexy depending upon their clinical evaluation. The participants will then be randomized to Restorelle® sacrocolpopexy
  Interventions: Device: Restorelle® Y mesh; Procedure: Laparoscopic sacrocolpopexy; Procedure: Robotic assisted laparoscopic sacrocolpopexy
- Vertessa® Lite Y mesh (Experimental): All subjects will be predetermined by their surgeon to undergo either a laparoscopic or robotic assisted laparoscopic sacrocolpopexy depending upon their clinical evaluation. The participants will then be randomized to Vertessa® Y sacrocolpopexy
  Interventions: Device: Vertessa® Lite Y mesh; Procedure: Laparoscopic sacrocolpopexy; Procedure: Robotic assisted laparoscopic sacrocolpopexy

INTERVENTIONS:
Device: Vertessa® Lite Y mesh — Via randomization, 50 surgical subjects will receive Vertessa® lite Y mesh for the treatment of vaginal vault prolapse. The patient will be blinded as to which mesh they receive.
  Arms: Vertessa® Lite Y mesh
Device: Restorelle® Y mesh — Via randomization, 50 surgical subjects will receive Restorelle® Y mesh for the treatment of vaginal vault prolapse.The patient will be blinded as to which mesh they receive.
  Arms: Restorelle® Y mesh
Procedure: Laparoscopic sacrocolpopexy — The subject's surgeon will decide if their patient should have laparoscopic sacrocolpopexy upon their clinical evaluation
Procedure: Robotic assisted laparoscopic sacrocolpopexy — The subject's surgeon will decide if their patient should have robotic assisted laparoscopic sacrocolpopexy upon their clinical evaluation

SUMMARY:
This is a randomized clinical trial to compare outcomes between the Restorelle® Y mesh and Vertessa® lite Y mesh for the treatment of vaginal vault prolapse.

Hypothesis: Vertessa® lite Y mesh is not inferior to Restorelle® Y mesh for the treatment of vaginal vault prolapse

DETAILED DESCRIPTION:
This is a randomized single-blind, non-inferiorty trial. Abdominal sacrocolpopexy is considered the gold standard for vault prolapse, and has demonstrated superior anatomic outcomes compared to transvaginal suspension procedures. Sacrocolpopexy involves suspension of the vagina to the anterior longitudinal ligament of the sacrum at the level of S1 using a bridging graft which can be made of biologic or synthetic materials. The graft is sutured to the anterior as well as the posterior vagina and then attached to the anterior longitudinal ligament of the sacrum. ). Both the Restorelle® Smartmesh (Coloplast, Inc., Minneapolis, MN, USA) and the Vertessa® lite mesh (Caldera Medical. Inc., Agoura Hills, CA, USA) are ultra-light macroporous polypropylene mesh grafts that are intended for pelvic floor reconstruction, both types of grafts are used to perform sacrocolpopexy. Currently no prospective data exists on the Vertessa® lite mesh for sacrocolpopexy. It is used by many surgeons, but there are no data showing that it is as efficacious in treating prolapse and avoiding mesh erosion in those patients undergoing sacrocolpopexy. Therefore, the primary objective of the proposed study is to compare outcomes between the Restorelle® Y mesh and Vertessa® lite Y mesh at the time of laparoscopic and robotic-assisted laparoscopic sacrocolpopexy.

Study subjects will be recruited from patients that present to the Center for Urogynecology & Pelvic Reconstructive Surgery in the Department of Obstetrics and Gynecology at the Cleveland Clinic Main campus, Hillcrest Hospital and Fairview Hospital, and their surgeries will be performed at either one of these sites. All subjects will be predetermined by their surgeon to undergo either a laparoscopic or robotic assisted laparoscopic sacrocolpopexy depending upon their clinical evaluation. The subjects will then we randomized to either Restorelle® or Vertessa® Y sacrocolpopexy according to a computer-generated randomization schedule with random block sizes with the use of the SAS statistical software package (SAS Institute, Cary, NC). All patients will be blinded to their assignment.

All subjects will be seen at a preoperative visit, then again at 6, 12 and 24 months postoperatively. During each visit. a vaginal exam and a complete Pelvic Organ Prolapse Quantification (POP-Q) exam will be performed. In addition, patients will be asked to complete the Pelvic Floor Distress Inventory (PFDI-20), Incontinence Severity Index (ISI) and Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) questionnaires at the preoperative visit as well as the 6, 12, and 24 month postoperative visits.

Laparoscopic sacrocolpopexy will be performed using four ports: an umbilical port for the laparoscope, two ports (either 5 or 10/12 mm) in the bilateral lower quadrants, and one 5-mm port placed at the level of the umbilicus, lateral to the rectus muscle on either side for retraction. The robotic-assisted hysterectomy will be performed using the da Vinci Surgical System (Intuitive Surgical Inc., Sunnyvale, CA, USA) using five ports: a 12mm umbilical port for the laparoscopic, two 8 mm robotic ports placed 2cm inferior and 9-10cm lateral to the umbilicus bilaterally, an 8mm robotic port placed in the left axillary line at the level of the umbilicus, and a 8mm or 10/12mm accessory port either in the right upper quadrant approximately 3cm distal from the costal margin, or in the right lower quadrant, 2cm above and medial to the anterior superior iliac spine.

If a supracervical hysterectomy is to be performed, it will be done in a standard fashion. A uterine manipulator will be placed inside of the uterus. The round ligaments will be transected using cautery. The fallopian tubes and ovaries will be left in situ or removed at the time of hysterectomy depending upon the preoperative decision made between the surgeon and patient. The uterine arteries and cardinal ligaments will be cauterized laparoscopically. The uterus will be amputated at the level of the internal cervical os and the endocervical canal will be cauterized.

The sacrocolpopexy will also be performed and in a standard fashion. An end-to-end anastomosis (EEA) sizer will be placed in the vagina for manipulation of the apex as well as in the rectum for delineation of the rectovaginal septum. First, the presacral dissection will be performed with a longitudinal peritoneal incision over the sacral promontory and there is identification of the anterior longitudinal ligament. Dissection is then done caudally through the peritoneum and subperitoneal fat down to the level of the posterior cul-de-sac. The vagina is elevated cephalad using the EEA sizer and the peritoneum overlying the anterior vaginal apex is incised transversely, and the bladder is dissected off the anterior vagina using sharp dissection, creating a 4 to 5 cm pocket. If this plane is difficult to establish, the bladder will be filled in a retrograde fashion to find the correct dissection plane. Similarly, the peritoneum overlying the posterior vagina is incised, and dissection is then done overlying the vagina and extending into the posterior cul-de-sac, creating a 4 to 5 cm pocket. Once dissection is complete, the mesh graft is prepared. Subjects will have been randomized to either one of two mesh grafts:

The Y mesh is introduced into the pelvis through one of the ports. First, either then anterior or the posterior arm is fixed to the anterior or posterior vaginal wall using 6 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other. The opposing arm of the graft is then attached to either the anterior or posterior vaginal wall, depending on which arm was placed first, in a similar fashion using 6 delayed- absorbable (PDS) No. 2-0 sutures in an interrupted fashion, 1 to 2 cm apart from each other. The stem portion of the graft is then brought to the sacral promontory and sutured to the anterior longitudinal ligament using 2 permanent (prolene) No. 0 sutures. The excess mesh is then trimmed.

The peritoneum is then closed over the exposed graft with absorbable suture. Routine cystoscopy will also be performed in order to assess for lower urinary tract injury. A vaginal exam is performed, and an anterior and/or posterior colporrhaphy and perineorrhaphy are performed if needed. Anti-incontinence procedures may also be performed if needed.

Preoperative data will include the following:

* Patient age, race, vaginal parity, menopausal sate, BMI, prior prolapse surgery, preoperative prolapse stage
* PFDI-20, ISI, PISQ-12
* Preoperative hemoglobin

Data points recorded during the procedure will include:

* Total OR time = operating room time of entry and exit
* Total Case time = time from incision to closure
* Concomitant procedures

  * Supracervical hysterectomy
  * Anterior colporrhaphy
  * Posterior colporrhaphy
  * Perineorrhaphy
  * Midurethral sling
* Estimated blood loss
* Intraoperative complications

  * EBL > 500cc
  * Vascular Injury
  * Cystotomy
  * Ureteral Injury
  * Bowel Injury - small bowel, large bowel, rectal

Postoperative data will include the following: 6, 12, 24 months

* POP-Q exam (performed by a provider blinded to the mesh used at the time of the procedure)
* PFDI-20, ISI, PISQ-12
* Review of electronic medical record (inpatient notes, d/c summary, ER visits), assessing for postoperative complications

  * Reoperation for immediate complications = reoperation within 30 days of surgery
  * Abdominal Wound infection = fascial, subcutaneous, cutaneous infection requiring antibiotic treatment
  * Hematoma = intrapelvic/abdominal
  * Vaginal cuff cellulitis/Pelvic Abscess = requiring IV/PO antibiotic therapy and/or transvaginal, trangluteal or percutaneous drainage
  * DVT/PE = diagnosed with Doppler US or CT scan
  * Reoperation for SUI with pubovaginal sling (synthetic or fascial), colposuspension, injection with periurethral bulking agents
  * Reoperation for mesh exposure
  * Reoperation for recurrent POP
  * Bowel Injury/Bowel Obstruction = enterotomy, perforation, ileus, partial/complete obstruction
  * Port site or incisional hernia
  * Need for any radiologic imaging
  * Lower urinary tract injury = bladder, ureteral
  * Neurologic Injury = brachial plexus, abdominal wall (ilioinguinal, iliohypogastric), lower extremity (femoral, sciatic, common peroneal)
  * Pulmonary complications = pneumonia, pulmonary hypertension, pulmonary edema within 14 days of surgery
  * Cardiac = ACS, MI, HF within 14 days of surgery
  * Postoperative ICU admission

Protection of each subject's personal health information will be a priority in this study. One master excel file containing subject personal information including name and medical record number will be kept in a password-protected file, on a designated protected research drive on a password-protected computer in a locked office at the Cleveland Clinic. In that file, each subject will be assigned a subject identification number that will be used for the purposes of data collection in order to de-identify subjects.

All paper forms used for data collection will be kept in a research cabinet dedicated to this project which will be locked at all times, in a locked office at the Cleveland Clinic. All forms will contain de-identified information - identification numbers will correspond to the subjects listed in the master excel file.

All study data will be transferred and managed electronically using REDCap (Research Electronic Data Capture). Each subject will be entered into REDCap using the assigned identification number from the master excel file. REDCap is a secure, web-based application designed to support data capture for research studies, providing user-friendly web-based case report forms, real-time data entry validation, audit trials, and a de-identified data export mechanism to common statistical packages. They system was developed by a multi-institutional consortium which was initiated at Vanderbilt University and includes the Cleveland Clinic. The database is hosted at the Cleveland Clinic Research Datacenter in the JJN basement and is managed by the Quantitative Health Sciences Department. The system is protected by a login and Secure Sockets Layers (SSL) encryption. Data collection is customized for each study as based on a study-specific data dictionary defined by the research team with guidance from the REDCap administrator in Quantitative Health Sciences at the Cleveland Clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, who are to undergo laparoscopic or robotic laparoscopic sacrocolpopexy for pelvic organ prolapse
* Other concomitant laparoscopic or prolapse and anti-incontinence procedures (e.g., laparoscopic supracervical hysterectomy, cystocele repair, rectocele repair or mid-urethral sling procedures) will be performed at the primary surgeon's discretion.

Exclusion Criteria:

* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Medical illness precluding laparoscopy
* Need for concomitant surgeries not related to pelvic organ prolapse or incontinence
* Sacrocolpoperineopexy
* Need for dual flat mesh for sacrocolpopexy procedure (determined by surgeon)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A Unger, MD, MPH, Principal Investigator — Assistant Professor of Surgery. Center for Urogynecology and Pelvic Reconstructive Surgery; Obstetrics/Gynecology and Women's Health Institute, Cleveland Clinic, Cleveland OH; Marie Fidela R Paraiso, MD, Principal Investigator — Professor, Section Head of the Center for Urogynecology and Pelvic Reconstructive Surgery; Obstetrics/Gynecology and Women's Health Institute, Cleveland Clinic, Cleveland OH
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ganatra AM, Rozet F, Sanchez-Salas R, Barret E, Galiano M, Cathelineau X, Vallancien G. The current status of laparoscopic sacrocolpopexy: a review. Eur Urol. 2009 May;55(5):1089-103. doi: 10.1016/j.eururo.2009.01.048. Epub 2009 Feb 4. PMID 19201521
- [Background] Walters MD, Ridgeway BM. Surgical treatment of vaginal apex prolapse. Obstet Gynecol. 2013 Feb;121(2 Pt 1):354-374. doi: 10.1097/AOG.0b013e31827f415c. PMID 23344287
- [Background] Porges RF, Smilen SW. Long-term analysis of the surgical management of pelvic support defects. Am J Obstet Gynecol. 1994 Dec;171(6):1518-26; discussion 1526-8. doi: 10.1016/0002-9378(94)90395-6. PMID 7802061
- [Background] Birch C. The use of prosthetics in pelvic reconstructive surgery. Best Pract Res Clin Obstet Gynaecol. 2005 Dec;19(6):979-91. doi: 10.1016/j.bpobgyn.2005.08.013. Epub 2005 Sep 26. PMID 16185932
- [Background] Chu CC, Welch L. Characterization of morphologic and mechanical properties of surgical mesh fabrics. J Biomed Mater Res. 1985 Oct;19(8):903-16. doi: 10.1002/jbm.820190803. PMID 3880350
- [Background] Kaupp HA, Matulewicz TJ, Lattimer GL, Kremen JE, Celani VJ. Graft infection or graft reaction? Arch Surg. 1979 Dec;114(12):1419-22. doi: 10.1001/archsurg.1979.01370360073009. PMID 160778
- [Background] Salamon CG, Lewis C, Priestley J, Gurshumov E, Culligan PJ. Prospective study of an ultra-lightweight polypropylene Y mesh for robotic sacrocolpopexy. Int Urogynecol J. 2013 Aug;24(8):1371-5. doi: 10.1007/s00192-012-2021-7. Epub 2013 Jan 8. PMID 23296684

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Started | 54 | 52
Completed | 47 | 44
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (9) | 58 (10) | 60 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 52 | 106
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 52 | 106

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Pelvic Organ Prolapse Recurrence
Description: Retreatment for prolapse by either surgery or pessary
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
participants | 2 | 1

2. Secondary Outcome: Number of Participants With Postoperative Complications
Description: Any postoperative complication at 6 months, including the following:
  Wound Infection Hematoma Pelvic Abscess VTE/PE Bowel Injury, Bowel Obstruction Port Site Hernia Lower Urinary Tract Injury Neurologic Injury
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
participants | 0 | 2

3. Secondary Outcome: Number of Participants With Mesh Exposure
Description: Mesh exposure on physical exam up to 24 months following surgery
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
participants | 0 | 0

4. Secondary Outcome: Number of Participants With Stress Incontinence Retreatment
Description: Stress incontinence retreatment including urethral bulking or sling up to 24 months following surgery
Time Frame: 24 months
Measure: Number; unit: participants
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
participants | 2 | 2

5. Secondary Outcome: Mean Difference Between Baseline (Pre-procedure) and 24-months Post-procedure
Description: The PFDI-20 (Pelvic Floor Distress Inventory - 20 items) measures pelvic floor dysfunction symptoms across three scales (POPDI-6, UDI-6, CRADI-8), with each item scored 0-4; to score, sum items per scale, find the mean, then multiply by 25 (0-100 range), and add scale scores for a total PFDI-20 score (0-300), where higher scores mean worse distress. A score of 0 indicates no symptoms. Mild - less than or equal to 100; Moderate - greater than 100 but less than or equal to 200; and Severe - greater than 200.
Time Frame: Baseline (pre-procedure) to 24-months (post-procedure)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
units on a scale | -78.8 (49.8) | -75.1 (59.5)

6. Secondary Outcome: Mean Difference Between Baseline (Pre-procedure) and 24-months Post-procedure
Description: The Incontinence Severity Index (ISI) is a validated measure that quantifies urinary incontinence severity based on patient-reported frequency and amount of leakage. Scores are calculated by multiplying the frequency score (0-4) by the amount score (1-3), yielding possible total scores of 0, 1, 2, 3, 4, 6, 8, 9, and 12. The minimum possible score is 0, indicating no incontinence, and the maximum possible score is 12, indicating very severe incontinence. ISI scores are categorized as follows: 0 (dry), 1-2 (slight), 3-6 (moderate), 8-9 (severe), and 12 (very severe). Lower scores reflect less severe symptoms and represent more favorable outcomes, whereas higher scores indicate greater symptom burden and worse clinical outcomes. Improvement in incontinence severity is defined as a decrease in ISI score over time, while worsening is defined as an increase in score.
Time Frame: Baseline (pre-procedure) to 24-months (post-procedure)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
Number analyzed (Participants) | 47 | 44
units on a scale | -2.7 (6.1) | -1.3 (6.3)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Restorelle® Y Mesh | Vertessa® Lite Y Mesh
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 0/54 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT03681223/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/23/NCT03681223/ICF_001.pdf